CLINICAL TRIAL: NCT05482633
Title: Investigation of the Effects of Inspiratory Muscle Training on Respiratory Muscle Strength, Respiratory Functions and Aerobic Exercise Capacity in Children With Juvenile Idiopathic Arthritis: A Single-Blind Randomized Controlled Study
Brief Title: Inspiratory Muscle Training in Juvenile Idiopathic Arthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir Katip Celebi University (Other)
Responsible Party: Principal Investigator, Devrim Can Sarac, PhD(c), Research Assistant, Izmir Katip Celebi University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IMTJIA
Record Dates: First submitted 2022-07-01; First posted 2022-08-01 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Juvenile Idiopathic Arthritis
Keywords: Respiratory muscles; exercise; physiotherapy; respiratory muscle training
MeSH Terms: conditions — Arthritis, Juvenile; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: An independent assessor who is unaware of the group of participants going to perform all evaluations.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Experimental group is going to perform inspiratory muscle training exercises everyday for 8 weeks.
  Interventions: Other: Inspiratory muscle training (IMT)
- Control Group (No Intervention): No new interventions will be given to control group.

INTERVENTIONS:
Other: Inspiratory muscle training (IMT) — Treatment group will perform IMT every day for eight weeks. Initial load is going to be set as the 60% of maximal inspiratory pressure (PImax) and is going to be increased by %10 of the initial load every two weeks.
  Arms: Intervention Group

SUMMARY:
The aim of this study is to investigate the effectiveness of inspiratory muscle training (IMT) in increasing respiratory muscle strength in patients with juvenile idiopathic arthritis.

DETAILED DESCRIPTION:
Primary pulmonary involvement is an important aspect that leads to morbidity and mortality in adult patients with rheumatoid arthritis [1,2] but is not as frequent in patients with juvenile idiopathic arthritis (JIA), (prevalence; 4-8%) [3]. However, a body of evidence indicates that respiratory functions are affected in more than 50% of all children with JIA, even in those without radiological involvement [1,2,4]. Previous studies comparing children with JIA to their healthy peers showed that forced vital capacity (FVC), forced expiratory volume in 1 second (FEV1), peak flow rate (PEF), and carbon monoxide diffusion capacity (DLCO) are decreased and the maximum inspiratory pressure (PImax) and maximum expiratory pressures (PEmax), which are used to assess respiratory muscle strength, are significantly lower [2,4]. In addition, it has been reported that disease-modifying drugs (DMARDs) and non-steroidal anti-inflammatory drugs (NSAIDs), which are frequently used in the treatment of patients with JIA may cause a decrement in respiratory functions [5]. It has been suggested that the decrease in the pulmonary functions in patients with JIA without radiological involvement of the lung parenchyma or thorax may be caused by the weakness of inspiratory and expiratory muscles [2]. Moreover, symptoms and signs such as chronic joint pain and stiffness, synovitis, and deformity seen in children with JIA may limit movement, leading to an inactive lifestyle. Evidence suggests that children with JIA have lower levels of physical activity than age-matched controls [6,7]. This inactive lifestyle accompanying the disease process; may cause decline in aerobic and anaerobic capacity, peripheral muscle strength and quality of life [8,9].

Inspiratory muscle training (IMT) is defined as a technique that aims to improve the function and strength of respiratory muscles through performing exercises with a specialized device [10,11]. There is evidence that the IMT method improves functional status and increases respiratory muscle strength, respiratory volumes, and aerobic exercise capacity in adult rheumatologic patients [12,13]. IMT seems to increase perfusion and muscle metabolism in both respiratory and extremity muscles, provide muscle fiber type conversion, create neural plasticity at respiratory synapses in the central nervous system, and modulate dyspnea in different populations [14]. Despite this, the effectiveness of IMT has not been investigated in patients with JIA.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with JIA according to International League of Associations of Rheumatology (ILAR) criteria by a specialist pediatric rheumatologist.
* Being between the ages of 13-18.
* To be able to understand and speak the Turkish language adequately.
* Being on the same biological agent treatment for the last three months.
* Agreeing to participate in the research.
* The patient's family accepts the child's participation in the study.
* Having a history of arthritis in at least one joint in lower extremities.

Exclusion Criteria:

* Presence of a condition that prevents performing respiratory muscle training therapy
* Being involved in a different physiotherapy and rehabilitation program six months before the start of the study
* Having a regular exercise habit during last six months (applying a structured exercise program at least 3 days a week)
* Presence of a different pathology that may affect cardiovascular fitness, pulmonary capacity, walking capacity or quality of life.
* Being diagnosed with systemic JIA clinical subtype.

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 33 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2022-09-15 (Actual); Study Completion 2022-09-15 (Actual)

PRIMARY OUTCOMES:
Maximal inspiratory pressure (PImax) | Change from baseline PImax at 8th week
  Maximal inspiratory pressure (PImax) is the highest subatmospheric pressure achieved when inspiring against a closed airway.

SECONDARY OUTCOMES:
Maximal expiratory pressure (PEmax) | Change from baseline PEmax at 8th week
  Maximal expiratory pressure (PEmax) is the highest pressure achieved during forced expiration against a closed airway. PEmax is indicative of the strength of expiratory muscles.
Maximal Oxygen Consumption (VO2max) | Change from baseline VO2max at 8th week
  VO2max is going to be evaluated using Cardiopulmonary exercise test (CPET). CPET is a non-invasive procedure that evaluates an individual's capacity during dynamic exercise and provides diagnostic and prognostic information. CPET is based on the investigation of respiratory system, cardiovascular system and cellular response to exercise performed under controlled metabolic conditions.
Forced Vital Capacity (FVC) | Change from baseline FVC at 8th week
  FVC is going to be measured with spirometry. Spirometry is the most frequently used measure of lung function and is a measure of volume against time.
Forced Expiratory Volume in one second (FEV1) | Change from baseline FEV1 at 8th week
  FEV1 is going to be measured with spirometry. Spirometry is the most frequently used measure of lung function and is a measure of volume against time.

CONTACTS AND LOCATIONS:
Locations (1):
- Izmir Katip Celebi University, Izmir, Turkey (Türkiye)

REFERENCES:
- [Background] Richardson AE, Warrier K, Vyas H. Respiratory complications of the rheumatological diseases in childhood. Arch Dis Child. 2016 Aug;101(8):752-8. doi: 10.1136/archdischild-2014-306049. Epub 2016 Jan 14. PMID 26768831
- [Background] Alkady EA, Helmy HA, Mohamed-Hussein AA. Assessment of cardiac and pulmonary function in children with juvenile idiopathic arthritis. Rheumatol Int. 2012 Jan;32(1):39-46. doi: 10.1007/s00296-010-1548-5. Epub 2010 Jul 24. PMID 20658239
- [Background] Noyes BE, Albers GM, deMello DE, Rubin BK, Moore TL. Early onset of pulmonary parenchymal disease associated with juvenile rheumatoid arthritis. Pediatr Pulmonol. 1997 Dec;24(6):444-6. doi: 10.1002/(sici)1099-0496(199712)24:63.0.co;2-8. No abstract available. PMID 9448237
- [Background] Knook LM, de Kleer IM, van der Ent CK, van der Net JJ, Prakken BJ, Kuis W. Lung function abnormalities and respiratory muscle weakness in children with juvenile chronic arthritis. Eur Respir J. 1999 Sep;14(3):529-33. doi: 10.1034/j.1399-3003.1999.14c09.x. PMID 10543271
- [Background] Camiciottoli G, Trapani S, Castellani W, Ginanni R, Ermini M, Falcini F. Effect on lung function of methotrexate and non-steroid anti-inflammatory drugs in children with juvenile rheumatoid arthritis. Rheumatol Int. 1998;18(1):11-6. doi: 10.1007/s002960050047. PMID 9672993
- [Background] Henderson CJ, Lovell DJ, Specker BL, Campaigne BN. Physical activity in children with juvenile rheumatoid arthritis: quantification and evaluation. Arthritis Care Res. 1995 Jun;8(2):114-9. doi: 10.1002/art.1790080210. PMID 7794985
- [Background] Bohr AH, Nielsen S, Muller K, Karup Pedersen F, Andersen LB. Reduced physical activity in children and adolescents with Juvenile Idiopathic Arthritis despite satisfactory control of inflammation. Pediatr Rheumatol Online J. 2015 Dec 10;13:57. doi: 10.1186/s12969-015-0053-5. PMID 26653716
- [Background] van Brussel M, Lelieveld OT, van der Net J, Engelbert RH, Helders PJ, Takken T. Aerobic and anaerobic exercise capacity in children with juvenile idiopathic arthritis. Arthritis Rheum. 2007 Aug 15;57(6):891-7. doi: 10.1002/art.22893. PMID 17665476
- [Background] Bayraktar D, Savci S, Altug-Gucenmez O, Manci E, Makay B, Ilcin N, Unsal E. The effects of 8-week water-running program on exercise capacity in children with juvenile idiopathic arthritis: a controlled trial. Rheumatol Int. 2019 Jan;39(1):59-65. doi: 10.1007/s00296-018-4209-8. Epub 2018 Nov 14. PMID 30430201
- [Background] McConnell AK, Romer LM. Respiratory muscle training in healthy humans: resolving the controversy. Int J Sports Med. 2004 May;25(4):284-93. doi: 10.1055/s-2004-815827. PMID 15162248
- [Background] American Thoracic Society/European Respiratory Society. ATS/ERS Statement on respiratory muscle testing. Am J Respir Crit Care Med. 2002 Aug 15;166(4):518-624. doi: 10.1164/rccm.166.4.518. No abstract available. PMID 12186831
- [Background] Dragoi RG, Amaricai E, Dragoi M, Popoviciu H, Avram C. Inspiratory muscle training improves aerobic capacity and pulmonary function in patients with ankylosing spondylitis: a randomized controlled study. Clin Rehabil. 2016 Apr;30(4):340-6. doi: 10.1177/0269215515578292. Epub 2015 Mar 25. PMID 25810425
- [Background] Basakci Calik B, Gur Kabul E, Taskin H, Telli Atalay O, Bas Aslan U, Tasci M, Bicakci F, Yildiz AI. The efficiency of inspiratory muscle training in patients with ankylosing spondylitis. Rheumatol Int. 2018 Sep;38(9):1713-1720. doi: 10.1007/s00296-018-4093-2. Epub 2018 Jun 25. PMID 29943207
- [Background] Bissett B, Gosselink R, van Haren FMP. Respiratory Muscle Rehabilitation in Patients with Prolonged Mechanical Ventilation: A Targeted Approach. Crit Care. 2020 Mar 24;24(1):103. doi: 10.1186/s13054-020-2783-0. PMID 32204719